CLINICAL TRIAL: NCT06377826
Title: To Compare the Effects of Aerobic and Resistance Training on Exercise Capacity, Depression and Quality of Life in Hypothyroidism.
Brief Title: Comparison of Aerobic and Resistance Training on Exercise Capacity, Depression and Quality of Life in Hypothyroidism.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCRAHS-ISB/REC/MS-PT/01813
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Comparison of Aerobic Exercise and Resistance Training
MeSH Terms: interventions — Exercise; Resistance Training; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic exercises (Active Comparator): Aerobic exercises i-e treadmill walking, bicycle ergometer, Treadmill
  Interventions: Other: aerobic exercises
- resistance training (Experimental): resistance exercise training gluteal bridge, calf raises, squats, seated shoulder press,
  Interventions: Other: resistance training
- medication (Placebo Comparator): only on drugs no exercise is given
  Interventions: Drug: medication

INTERVENTIONS:
Other: aerobic exercises — group A will receive aerobic training like walking and cycling for 03 times per week approximately each exercise 5 to 10 minutes for 8 weeks.
  Arms: aerobic exercises
Other: resistance training — this group will receive resistance training like gluteal bridge, calf raise, squats, seated shoulder press for 03 times per week approximately each exercise 5 to 10 minutes for 8 weeks.
  Arms: resistance training
Drug: medication — This group will be just on medication and no exercise will be given to this group
  Arms: medication

SUMMARY:
the study will show the effects of aerobic and resistance training on exercise capacity, depression and quality of life in patients with hypothyroidism. The evaluation of TSH level before and after the exercise sessions will provide valuable data.

DETAILED DESCRIPTION:
The study aims to investigate the effects of aerobic exercise and resistance training by comparing the two types of exercises, the finding of this study gain insights into the most effective approach for patients with hypothyroidism particularly in relation to exercise capacity, depression and quality of life. The study design is Randomized Controlled Trial. Sample size is calculated using G power program. the study duration is 6 months after the approval of research board. Non probability Purposive sampling is used for this study. Data will be analyzed by using SPSS version 20.

ELIGIBILITY:
Inclusion Criteria:

Both males and females Age between 40 to 60 years Diagnosed cases of hypothyroidism Duration: 2 years being diagnosed Patients who easily perform exercises

Exclusion Criteria:

Patients with serious comorbidities like cancer Uncontrolled hypertension Vitally unstable patients Red flags for physiotherapy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test | 8 weeks
  The six minute walk test 96 The six minute walking test (6MWT) was developed by the American Thoracic Society and it was officially introduced in 2002, coming along with a comprehensive guideline. The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The 6-minute walk test (6MWT) is commonly used to measure the functional exercise capacity in chronic patients with cardiovascular disease.
The Beck Depression Inventory Scale | 8 weeks
  The Beck Depression Inventory (BDI, BDI-1A, BDI-II), created by Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Its development marked a shift among mental health professionals, who had until then, viewed depression from a psychodynamic perspective, instead of it being rooted in the patient's own thoughts. Each question had a set of at least four possible responses, ranging in intensity. Higher total scores indicate more severe depressive symptom.
SF- 36 SF-36 | 8 weeks
  SF- 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life.
  It comprises 36 questions that cover eight domains of health. The SF-36 is often used as a measure of a person or population's quality of life (QOL).

CONTACTS AND LOCATIONS:
Overall Officials: saira jahan, Principal Investigator — Riphah International University
Locations (1):
- Abbottabad medical complex, Abbottābād, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No